CLINICAL TRIAL: NCT00906100
Title: Prevalence of Prolonged Inter/Intra-Atrial Delay That Would Preclude Optimization of Atrioventricular (AV) Delay in Patients Undergoing Biventricular (BiV) Device Placement
Brief Title: Prevalence of Atrial Delay That Would Preclude Optimization of Atrioventricular (AV) Delay in Patients With Biventricular (BiV) Device
Status: Withdrawn | Type: Observational
Why Stopped: Dr Obel is deceased and no other investigators on study to provide information. old record, IRB has no information; outside of retention period.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Owen Obel, MD, UT Southwestern Medical Center
Other Study IDs: UTSW IRB 122007-040
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Biventricular ICD; AV delay
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the proportion of patients who are undergoing Biventricular (BiV) Implantable Cardioverter Defibrillator (ICD) implantation in whom optimization of atrioventricular (AV) delay is not possible due to prolonged inter-atrial/intra-atrial delay. These patients would benefit from left atrial pacing, and if a significant number of patients fall into this group, it may be beneficial to develop a left atrial lead.

DETAILED DESCRIPTION:
This is a prospective observational study. Patients referred for BiV-ICD implantation or upgrade will be implanted as is routinely done, with the following modifications:

* Electrical readings will be taken at various points in the procedure.
* The RA lead will temporarily be placed on the atrial septum for these readings (normally it is actively fixed to the RA appendage wall). The final RA lead position will be actively fixed to the RA appendage wall as is standard practice.
* The CS lead will be placed in the proximal coronary sinus for these readings prior to passing it distally to pace the LV.
* Patients will undergo transthoracic echocardiography (TTE) 30 days post-procedure. This will be coordinated to coincide with their standard 30-day follow-up appointment.

Conduction times between the left atrium and right atrium (inter-atrial conduction time) will be measured at the time of implant, and left atrial contraction time will be measured by TTE at the follow-up appointment. For patients in whom the inter-atrial conduction time plus the left atrial contraction time is greater than the right-atrial to right-ventricular conduction time, it is not possible to optimize the AV delay. The proportion of patients who fall into this group will be the main endpoint of the study. Patients will be followed for this study until their follow-up appointment and TTE at 30 days post-implant. The total sample size of this study will be 50 patients. We expect to consent approximately 75 patients, expecting that 1/3 will not meet all entrance criteria or will withdraw early.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Have the ability to provide informed consent and willingness to comply with follow-up tests
* QRS duration > 120 ms
* Ejection fraction < 35%
* Persistent symptoms of class III or IV heart failure despite a stable and optimized medical regimen
* Normal sinus rhythm or sinus bradycardia

Exclusion Criteria:

* White-Parkinson-White syndrome
* Chronic persistent atrial fibrillation
* Complete heart block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for biventricular ICD placement
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
to determine the proportion of patients who are undergoing Biventricular (BiV) Implantable Cardioverter Defibrillator (ICD) implantation in whom optimization of atrioventricular (AV) delay is not possible due to prolonged inter-atrial/intra-atrial delay.

CONTACTS AND LOCATIONS:
Overall Officials: Owen Obel, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States